CLINICAL TRIAL: NCT06269861
Title: Evaluation of the Relation of the Body Weight Calculated by Visual Estimation and Anthropometric Measurements to the Actual Body Weight Measured by the Patient Transfer Scale in Critically Ill Patients
Brief Title: Comparison of Body Weights Via Visual Estimation, Anthropometric Calculation, and Actual Measured in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nazlıhan Boyacı Dündar, assistant professor, Gazi University
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Screening
Other Study IDs: GaziUtipNBDundar003
Record Dates: First submitted 2024-02-10; First posted 2024-02-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Critically Ill; Body Weight
Keywords: actual body weight; ideal body weight; anthropometric measurements; patient transfer scale
MeSH Terms: conditions — Critical Illness; Body Weight

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: To avoid self-calibration, all measurements will be recorded by a different doctor other than the primary care physician.
  The all calculations will be performed by a different doctor other than the primary care physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- inward patients (Other): The inward patients who will be weighed with bathroom scale and patient transfer scale
  Interventions: Device: patient transfer scale
- critically ill patients (Other): The critically ill patients who will be weighed with patient transfer scale
  Interventions: Device: patient transfer scale

INTERVENTIONS:
Device: patient transfer scale — patient transfer scale is a device to measure actual weight for critically ill patient who are unable to stand

SUMMARY:
Rapid and accurate determination of body weight in adult intensive care patients is very important for both calculating target tidal volume during invasive mechanical ventilation support and dose dependent drug administration. In this patient group, measuring actual body weight with a calibrated scale by standing the patient up is often impossible due to acute illness. Instead, estimated body weight determined by health care personnel or estimated body weights calculated according to anthropometric measurements are used. These calculations have some limitations in showing actual body weight, and there is some controversial information in current literature regarding their validity in critically ill patients. There is newly developed patient transfer scale called Marsden M-999® manufactured by Marsden Weighing Machine Group Ltd, which has the advantage of being used in patients who are unable to stand up, in rapidly and accurately measuring the current body weight in critically ill patients. This study aimed to evaluate the validity of these methods by comparing the body weights calculated by visual estimation and various anthropometric methods in critically ill Turkish patients with the actual weight measured by the mentioned scale.

DETAILED DESCRIPTION:
In adult medicine, determining the patient's body weight by visual estimation performed by healthcare providers (nurses and doctors) is common for critically ill patients who cannot speak or stand due to acute illnesses such as loss of consciousness, circulatory shock, or acute respiratory failure. This practice often leads to the administration of the same dose of medication to many patients whose body weight may vary between 50 to 100 kilograms (kg). In cases where rapid diagnosis and treatment are crucial due to acute illness, the accurate and effective administration of dose-dependent drugs such as antibiotics, anticoagulants, vasopressors, sedatives, and analgesics is essential for treatment success. Although the average error percentage of 10-20% in estimated body weight by visual estimation may seem negligible in emergencies, it can lead to increased toxicity and costs in recombinant factor replacements, anticoagulants with a narrow therapeutic range, and various imported antibiotics. Additionally, the high error rate in estimating height by visual estimation poses a risk of causing ventilator-induced lung injury (VILI) during invasive mechanical ventilation support by inducing alveolar overdistension.

Various calculation methods have been reported for estimating body weight based on anthropometric measurements. One such method is weight calculation based on the upper mid-arm circumference (UMAC), which has been reported as the most correlated calculation for actual body weight in the adult age group in studies using National Health and Nutrition Examination Survey (NHANES) data in the United States (U.S.). Another commonly used method is formulas that calculate ideal body weight based on the patient's height. This is especially crucial in critically ill patients during invasive mechanical ventilation support for acute respiratory failure. The calculation of ideal body weight using charts based on half-span or knee height can be applied in cases where patients cannot stand due to critical illness.

Many anthropometric measurements mentioned here have been conducted in different societies. They may vary according to ethnic communities, emphasizing the potential differences in body composition, such as fat and muscle mass distribution, among different ethnic groups. Considering the critical illness in the Turkish population, there is currently no detailed publication in the literature regarding the usability of estimated body weights calculated based on anthropometric measurements. Moreover, the fact that many anthropometric measurements are derived from population screening data in healthy individuals causes their application in clinical practice challenging. Validity of anthropometric measurements that apply to critically ill patients, where patients cannot stand, appropriate positions for anthropometric measurements cannot be provided, and body distributions in limbs where anthropometric measurements are derived may differ due to peripheral edema, is, therefore, crucial.

In many studies using anthropometric measurements for weight calculation, the actual body weights of patients were measured using a calibrated scale. Given that critically ill patients often cannot be lifted due to acute illness, special devices or equipments are needed to reliably determine actual body weights in the supine position in this patient group. Currently, used bed scales, wall-mounted levers, or special devices that allow the patient and bed to be weighed together are not widely used due to high costs and difficulties associated with patient transfer from bed to bed, such as the need for the patient to be hemodynamically stable, the need for multiple personnel during patient transfer, adherence to infection prevention rules, and the time-consuming nature of measurements depending on the device used. The recently developed patient transfer scale, Marsden M-999®, which has advantages for patients who cannot stand, suggests that it could be used to calculate actual weight rapidly and accurately in critically ill patients. There is no publication currently in the literature about the routine use of the mentioned patient transfer scale in critically ill settings. However, its ease of use in measuring patient body weight in the supine position while transitioning from a stretcher to an intensive care bed is a significant advantage.

Considering that the patient transfer scale cannot be provided to every intensive care unit due to its cost; it was aimed to determine the most valid estimated body weight calculation method in the critically ill Turkish patients according to anthropometric measurements in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can stand without assistance are admitted to the inward of the internal disease department.
2. Patients who are admitted to the medical intensive care units

Exclusion Criteria:

1. Patient or control group under the age of 18 years
2. Patients died within the first 8 hours after hospital admission
3. Patients who did not sign informed consent
4. Refusal of legal representative to participate in the study in unconscious patients
5. Patients with anatomical defects or limb instruments that would prevent performing anthropometric measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
determining actual weight | Actual body weight measured with bathroom scales and patient transfer scales in standing patients on the day of hospital; up to 8 weeks for purpose of reaching total patients number of 100
  The correlation between actual weight measured with bathroom scales and patient transfer scales in standing patients
determining the ideal estimated body weight in critically ill patients | Actual and estimated weight of patients determined on the first day of intensive care unit; up to 6 months for purpose of reaching total patients number of 100
  The correlation of actual weight with estimated weight determined based on visual estimation and anthropometric measurements in critically ill

CONTACTS AND LOCATIONS:
Overall Officials: Nazlıhan Boyacı Dündar, asist. prof., Principal Investigator — Gazi University, Faculty of Medicine
Locations (1):
- Gazi University, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cattermole GN, Graham CA, Rainer TH. Mid-arm circumference can be used to estimate weight of adult and adolescent patients. Emerg Med J. 2017 Apr;34(4):231-236. doi: 10.1136/emermed-2015-205623. Epub 2016 Dec 19. PMID 27993936
- [Background] Maskin LP, Attie S, Setten M, Rodriguez PO, Bonelli I, Stryjewski ME, Valentini R. Accuracy of weight and height estimation in an intensive care unit. Anaesth Intensive Care. 2010 Sep;38(5):930-4. doi: 10.1177/0310057X1003800519. PMID 20865881
- [Background] Bloomfield R, Steel E, MacLennan G, Noble DW. Accuracy of weight and height estimation in an intensive care unit: Implications for clinical practice and research. Crit Care Med. 2006 Aug;34(8):2153-7. doi: 10.1097/01.CCM.0000229145.04482.93. PMID 16763505
- [Background] Breuer L, Nowe T, Huttner HB, Blinzler C, Kollmar R, Schellinger PD, Schwab S, Kohrmann M. Weight approximation in stroke before thrombolysis: the WAIST-Study: a prospective observational "dose-finding" study. Stroke. 2010 Dec;41(12):2867-71. doi: 10.1161/STROKEAHA.110.578062. Epub 2010 Nov 11. PMID 21071723
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Venkataraman R, Ranganathan L, Nirmal V, Kameshwaran J, Sheela CV, Renuka MV, Ramakrishnan N. Height measurement in the critically ill patient: A tall order in the critical care unit. Indian J Crit Care Med. 2015 Nov;19(11):665-8. doi: 10.4103/0972-5229.169342. PMID 26730118
- [Background] L'her E, Martin-Babau J, Lellouche F. Accuracy of height estimation and tidal volume setting using anthropometric formulas in an ICU Caucasian population. Ann Intensive Care. 2016 Dec;6(1):55. doi: 10.1186/s13613-016-0154-4. Epub 2016 Jun 21. PMID 27325410
- [Background] Hickson M, Frost G. A comparison of three methods for estimating height in the acutely ill elderly population. J Hum Nutr Diet. 2003 Feb;16(1):13-20. doi: 10.1046/j.1365-277x.2003.00416.x. PMID 12581405
- [Background] Bassey EJ. Demi-span as a measure of skeletal size. Ann Hum Biol. 1986 Sep-Oct;13(5):499-502. doi: 10.1080/03014468600008661. PMID 3800311
- [Background] Chumlea WC, Guo S, Roche AF, Steinbaugh ML. Prediction of body weight for the nonambulatory elderly from anthropometry. J Am Diet Assoc. 1988 May;88(5):564-8. PMID 3367012
- [Background] Opdam MH, Koekkoek KWAC, Boeije T, Mullaart N, van Zanten ARH. Mid-arm circumference method is invalid to estimate the body weight of elderly Emergency Department patients in the Netherlands. Medicine (Baltimore). 2019 Aug;98(32):e16722. doi: 10.1097/MD.0000000000016722. PMID 31393379
- [Background] Kokong DD, Pam IC, Zoakah AI, Danbauchi SS, Mador ES, Mandong BM. Estimation of weight in adults from height: a novel option for a quick bedside technique. Int J Emerg Med. 2018 Nov 27;11(1):54. doi: 10.1186/s12245-018-0212-9. PMID 31179934
- [Background] Freitag E, Edgecombe G, Baldwin I, Cottier B, Heland M. Determination of body weight and height measurement for critically ill patients admitted to the intensive care unit: A quality improvement project. Aust Crit Care. 2010 Nov;23(4):197-207. doi: 10.1016/j.aucc.2010.04.003. Epub 2010 Jun 25. PMID 20576445